CLINICAL TRIAL: NCT02044497
Title: Population Pharmacokinetics and Pharmacogenomics of Oral Oxycodone in Pediatric Surgical Patients
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Patcharee Sriswasdi, MD, Boston Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB-P00006691
Record Dates: First submitted 2014-01-22; First posted 2014-01-24 (Estimated); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Pediatric Surgical Patient
Keywords: pharmacokinetics; pharmacogenomics; oral oxycodone; pediatric surgical patients
MeSH Terms: interventions — Oxycodone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- oral oxycodone (Experimental): An orogastric tube will be placed in the stomach (placement verified by routine accepted clinical guidelines) under anesthesia as is part of standard routine clinical care to remove gastric contents. The same orogastric tube will be used for intragastric liquid oxycodone administration in a dose of 0.1 mg/kg before the surgical incision. This weight-adjusted dose of 0.1 mg/kg is administered as per standard clinical dosing guidelines at Boston Children's Hospital.
  Interventions: Drug: oral oxycodone

INTERVENTIONS:
Drug: oral oxycodone

SUMMARY:
Oxycodone is an oral opioid analgesic that is most commonly prescribed for the management of pain in post-operative patients at Boston Children's Hospital. Oxycodone has been widely used in adults and children to relieve post-operative pain. However, its pharmacokinetics (what it does in the body) and pharmacodynamics (how it works) have not been well established in children. Some children, because of their specific genetic make-up, may metabolize the drug more quickly and therefore may be at risk for more side effects in the commonly prescribed dose. We would like to find out more about how this drug is absorbed, metabolized and excreted in children. In order to study these aspects, we would like to give oxycodone to surgical patients at Boston Children's Hospital then measure its metabolic activity and also perform a genetic analysis. The genetic testing is specifically to analyze the following genotypes only: cytochrome P450 2D6 (CYP2D6) and cytochrome P450 3A4 (CYP3A4), which represent the differences in cytochrome P450 metabolism of oxycodone.

DETAILED DESCRIPTION:
Oxycodone is the most commonly used analgesic for the management of moderate and severe postoperative pain. The efficacy of Oxycodone as a potent opioid has been confirmed in children.

The principal metabolic pathway of oxycodone in humans is N-demethylation via enzyme CYP3A4 to generate inactive noroxycodone. [6] A smaller amount (approximately 11%) is O-demethylated by cytochrome P450 enzyme CYP2D6 to become oxymorphone, the active and potent metabolite which exhibits about 40 times the affinity and 8 times the potency on μ-opioid receptors compared to the mother substance. Approximate frequencies of cytochrome P450 enzyme CYP2D6 phenotypes for the Caucasian population are: poor metabolizers 5 - 10%, extensive/intermediate metabolizers 65-90%, and ultra-rapid metabolizers 5 - 10%. Kirchheiner and colleagues noticed more codeine-related sedative side-effects in ultra-rapid metabolizers. In studies investigating extensive and poor metabolizers, codeine side-effects do not seem to be related to CYP2D6 genotype. However, clinical investigations of CYP2D6 genotype in the postoperative pain setting have shown conflicting results, and well-designed prospective studies are lacking. Taken together, these results demonstrate the need for careful pharmacokinetic studies in children who received a pharmacologic agent, such as oxycodone, which is metabolized by the enzyme CYP2D6.

The population PK of oxycodone and its metabolites has not been fully established for oral oxycodone in pediatric patients. In addition, there is a group of ultra-rapid metabolizers (approximately 4.5% of the population, but as high as 20% in some particular ethnic groups; East African and Saudi Arabian populations) which may be at risk for serious side effects in the commonly prescribed dose (which is extrapolated from adult recommendations). Given that BCH has switched (from codeine) to oxycodone as the most common opioid prescribed for all postoperative patients and the recent concerns of serious side effects from codeine. It is important to further investigate oral oxycodone to optimize dosing recommendations.

ELIGIBILITY:
Inclusion Criteria:

* A total of 68 generally healthy, opioid-naive children, aged 0-6 years, scheduled as in-patient surgery for ventriculoperitoneal shunt placement/revision or Craniotomy (Neurosurgery service), Cleft lip/palate repair (plastic surgery service) and hypospadias repair or ureteral urethral reimplantation (genitourinary surgery service) will be enrolled in the study.

Exclusion Criteria:

* Children will be excluded if they are currently taking any medications which are CYP3A4 or CYP2D6 inhibitors/inducers or have a history of allergy or hypersensitivity to oxycodone, have any condition that might interfere with GI absorption, distribution, hepatic metabolism or renal excretion of r oxycodone, or a diagnosis of sleep apnea or impaired respiratory reserve.

Max Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 68 (Estimated)
Dates: Start 2014-05; Primary Completion 2026-05 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Oxycodone, oxymorphone, noroxymorphone and noroxycodone serum levels | The 10 samples will be drawn at the following time points: 8 blood samples will be taken at 30 minutes, 1, 1.5, 2, 3, 4, 5, and 6 hours post-dose in every patient along other 2 samples at approximately either 8 and 12 or 10 and 24 hours post-dose.
  Oxycodone, oxymorphone, noroxymorphone and noroxycodone levels, at 10 time points, will be used to determine the single-dose Pharmacokinetics (PK) metric.

CONTACTS AND LOCATIONS:
Overall Officials: Patcharee Sriswasdi, MD, Principal Investigator — Boston Children Hospital
Locations (1):
- Boston Children Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided
Still formulating.